CLINICAL TRIAL: NCT03483740
Title: Cognitive Remediation Group Therapy to Improve Older Adults' Ability to Cope With HIV-Associated Neurocognitive Disorder (HAND)
Brief Title: Psychosocial Intervention for Older HIV+ Adults With HAND
Acronym: IN-HAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: CIHR Canadian HIV Trials Network (Network); Unity Health Toronto (Other); AIDS Committee of Toronto (Other); Factor-Inwentash Faculty of Social Work, University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CTNPT 029
Record Dates: First submitted 2018-01-09; First posted 2018-03-30 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2022-11

CONDITIONS: HIV/AIDS; Aging; Mild Cognitive Impairment; Group, Peer
Keywords: HIV-Associated Neurocognitive Disorder (HAND); Cognitive remediation group therapy; Mutual aid group therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This is a pilot, parallel design, randomized, controlled trial (RCT) that will allocate a sample (n=16) of people (≥ 40 yrs old) aging with HIV who have been diagnosed with MND from St. Michael's Hospital (SMH) in Toronto to either arm 1: 8 weekly 3-hour sessions of CRGT; or arm 2: 8 weekly 3-hour sessions of HIV group therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive remediation group therapy (Experimental): 8 weekly 3-hour sessions of CRGT
  Interventions: Behavioral: CRGT
- Mutual aid support group (Active Comparator): 8 weekly 3-hour sessions of HIV group therapy
  Interventions: Behavioral: HIV group therapy

INTERVENTIONS:
Behavioral: CRGT — Cognitive remediation group therapy (CRGT) will be comprised of 1/3 brain training exercises on tablets using PositScience software by BrainHQ and 2/3 mindfulness-based stress reduction (MBSR) involving various activities such as meditation, breathing exercises, etc. Intervention will comprise of 8 weekly 3-hour sessions.
  Arms: Cognitive remediation group therapy
Behavioral: HIV group therapy — These groups use a model of mutual aid to encourage peer-based discussion on the effects of living with HIV. Topics are determined by the group; facilitators ensure that safety is maintained throughout and make connections between participants as appropriate. Intervension will comprise of 8 weekly 3-hour sessions.
  Arms: Mutual aid support group

SUMMARY:
CTNPT 029 will test the feasibility and acceptability of cognitive remediation group therapy in older adults living with HIV who have been diagnosed with HIV-associated neurocognitive disorder (HAND). The cognitive remediation therapy will include tablet-based cognitive training and mindfulness-based stress reduction sessions.

DETAILED DESCRIPTION:
Approximately half of the aging HIV-positive population will be affected by HAND, making cognitive impairment related to HIV a significant comorbidity in this population. With the development, access to, and early initiation of modern antiretroviral therapy (ART), HAND is less severe and less common than it once was. However, people who were treated with old therapies, ones that were less effective and with higher rates of toxicity compared to current regimens, or who experienced AIDS defining illnesses, may be affected by HAND more frequently and more severely. Issues with cognition, memory, processing new information, problem solving, and decision making are all potential symptoms.

Psychosocial interventions have been used to decrease stress and depression and improve coping and quality of life in the general aging population experiencing cognitive impairment and depression. These techniques, which can vary widely, have not been fully tested in people aging with HAND.

CTNPT 029 (a pilot trial funded by the CTN) seeks to enroll 16 people at St. Michael's Hospital in Toronto. Study participants will be randomized to either receive cognitive remediation group therapy (CRGT) or standard HIV group therapy (control group). Both group therapies consist of a series of weekly 3-hour sessions led by a certified social worker and a peer. The CRGT group will spend one hour per session on brain training exercises (PositScience Software) and the remaining two hours on mindfulness-based stress reduction (meditation, breathing exercises, etc.). The control group will focus on general health and wellbeing for people aging with HIV. Study investigators will determine the usefulness of the structure of the sessions and the feasibility and acceptability of performing a study of this kind.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female; aged ≥ 40 years
2. Documented HAND diagnosis of Mild Neurocognitive Disorder (MND)
3. ≥ 5 years of HIV infection
4. Provided consent to St. Michael's Hospital to be contacted for future research studies
5. Can feasibly attend 8 weeks of group therapy in downtown Toronto

Exclusion Criteria:

1. Documented HAND diagnosis of asymptomatic neurocognitive impairment (ANI) or HIV-associated dementia (HAD)
2. Hospitalization within past 1 month
3. Inability to communicate in English
4. Inability to use a tablet
5. Anyone deemed by the principal investigator to be disruptive to a support group setting

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Walmsley, MD, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - AIDS Committee of Toronto (ACT), Toronto, Ontario
  - St. Michael's Hospital Neurobehavioral Research Unit, Toronto, Ontario
  - University Health Network, Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eaton AD, Walmsley SL, Craig SL, Rourke SB, Sota T, McCullagh JW, Fallon BA. Protocol for a pilot randomised controlled trial evaluating feasibility and acceptability of cognitive remediation group therapy compared with mutual aid group therapy for people ageing with HIV-associated neurocognitive disorder (HAND) in Toronto, Canada. BMJ Open. 2019 Oct 31;9(10):e033183. doi: 10.1136/bmjopen-2019-033183. PMID 31676660

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Remediation Group Therapy | Mutual Aid Support Group
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Remediation Group Therapy | Mutual Aid Support Group | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (6.72) | 59.7 (10.63) | 55.6 (8.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 4 | 9
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - Session Attendance
Description: Number of Participants who Attended at least 80% of the Group Sessions.
Time Frame: Three months
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Remediation Group Therapy | Mutual Aid Support Group
Number analyzed (Participants) | 6 | 6
Participants | 5 | 5

2. Primary Outcome: Acceptability - Participant Satisfaction With Group Sessions
Description: Participants will complete the Helping Characteristics of Self-Help and Support Groups Measure that will be complemented by questions about session length, number of sessions, activities used, and evaluation of facilitators.
  The Helping Characteristics of Self-Help and Support Group Measure contains 22 items that are scored on a 5-point-Likert style scale for a minimum score of 22 and a maximum score of 110. Higher scores indicate better outcome (outcome being satisfaction with support group). There are no subscales.
Time Frame: Three months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Cognitive Remediation Group Therapy | Mutual Aid Support Group
Number analyzed (Participants) | 6 | 6
score on a scale | 90 [74 to 100] | 85 [58 to 100]

3. Other Pre Specified Outcome: Change in Stress
Description: Assessed by the 'HIV/AIDS Stress Scale' at three time points. Score from 0 to 116. Lower scores mean better outcomes.
Time Frame: Baseline visit (week -1), follow-up visit (week 9), and end of study visit (week 21)
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Sustained Use of Brain Training Activities
Description: Self-report at three time points
Time Frame: Baseline visit (week -1), follow-up visit (week 9), and end of study visit (week 21)
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Sustained Use of Mindfulness Strategies
Description: Assessed by the 'Five Facet Mindfulness Questionnaire - Short Form' at three time points. Score from 24 to 120. Higher scores mean better outcomes.
Time Frame: Baseline visit (week -1), follow-up visit (week 9), and end of study visit (week 21). Score from 0 to 26
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Anxiety
Description: Assessed by the 'Anxiety in Cognitive Impairment and Dementia Scale' at three time points. Score from 0 to 26. Lower scores mean better outcomes.
Time Frame: Baseline visit (week -1), follow-up visit (week 9), and end of study visit (week 21)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Coping
Description: Assessed by the 'Coping Self-Efficacy Scale of Health Problems' at three time points. Score from 0 to 30. Higher scores mean better outcomes.
Time Frame: Baseline visit (week -1), follow-up visit (week 9), and end of study visit (week 21)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cognitive Remediation Group Therapy | Mutual Aid Support Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/40/NCT03483740/Prot_SAP_002.pdf
  • Informed Consent Form (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/40/NCT03483740/ICF_001.pdf